CLINICAL TRIAL: NCT04241432
Title: Acute Bone Response to Vibration in Boys Who Have a History of Fracture
Brief Title: Vibration in Boys With a History of Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SCH/11/061
Record Dates: First submitted 2018-04-18; First posted 2020-01-27 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Fracture
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Platform type 1 (Active Comparator): 12 pre-pubertal boys, aged 9-12 years who have previously sustained at least one fracture.
  Interventions: Device: vibrating platform
- Platform type 2 (Active Comparator): 12 pre-pubertal boys, aged 9-12 years who have previously sustained at least one fracture.
  Interventions: Device: vibrating platform

INTERVENTIONS:
Device: vibrating platform — Use of two different types of vibrating platform

SUMMARY:
Boys aged 9-12 years, with a history of facture will be asked to stand on one of two vibrating platforms for 10 minutes on 5 consecutive days. The investigators will take blood samples before and after the vibration to measure changes in the bone cells.

DETAILED DESCRIPTION:
Fractures in children are common, accounting for 10% of attendances in Accident and Emergency Departments. Research into risk factors for fracture has found that children who have narrower bones and a low bone mass are more likely to fracture than children with larger bones. Studies in postmenopausal women, young women with low bone mass and children with disabling conditions such as cerebral palsy, have shown that up to 10 minutes a day stood on a vibrating platform can significantly increase bone mass.

However little is known of the immediate response of bone to whole body vibration (WBV). The investigators previously investigated the acute bone response in healthy pre-pubertal boys to standing on one of two vibrating platforms for 10 minutes on 1, 3 or 5 consecutive days. This showed a platform dependent reduction in the bone resorption marker CTx pre to post vibration, with an increase in the bone formation marker P1NP over the 8 day study. The investigators would like to look at the response of bone to WBV in pre-pubertal boys who have a history of fracture(s). The investigators will compare this to the investigator's previous data to determine if bone in boys who have previously fractured responds in the same way as bone in boys who have not.

The investigators plan to recruit 24 boys aged 9-12 years who have had a previous fracture to stand on one of two vibrating platforms for 10 minutes on 5 consecutive days. Before and after the period of vibration on days 1, 3, 5, and on days 8 and 12 the investigators will take a blood sample to measure changes in the bone cells. The boys will be asked about the amount of exercise they have participated in over the previous seven days. The findings of this study will be used to direct further research.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Aged 7-13yrs (pre-pubertal)
* First language English
* History of one or more fracture(s)

Exclusion Criteria:

* Pre-existing chronic illness
* Known bone disease
* Current or healing fracture
* Recent (last 12 months) or current treatment likely to affect bone - this does not include inhaled or intermittent oral therapy with steroids for asthma
* Balance problems
* Continuing involvement in more than one other research study

Ages: 7 Years to 13 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2012-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Serum bone turnover marker concentrations: P1NP and CTX (ng/ml) | 68 months
  Serum bone turnover marker concentrations: P1NP and CTX (ng/ml)
Serum bone factor concentrations: OPG and sclerostin (pg/ml) | 68 months
  Serum bone factor concentrations: OPG and sclerostin (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Harrison, Principal Investigator — Investigator
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, Sheffield (South Yorkshire District), United Kingdom

IPD SHARING:
Plan to Share IPD: No